CLINICAL TRIAL: NCT03469986
Title: Prospective, Pivotal, Double-Blinded Within-subject Comparison of the Marcus Autism Center Investigational Device and Current Best Practice Clinical Diagnosis For Autism Spectrum Disorder in Pediatric Subjects 16-30 Months of Age
Brief Title: A Multi-site Comparison of Social Visual Engagement to Clinical Diagnosis for Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: EarliTec Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: S-DTD-2014-301
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: Children who meet criteria based on expert clinical diagnosis for autism spectrum disorder will be tested with the Marcus Autism Center Investigational Device and expert clinical assessment.
  Interventions: Device: Marcus Autism Center Investigational Device
- Non-autism Spectrum Disorder: Children who do not meet criteria for autism spectrum disorder based on expert clinical diagnosis will be tested with the Marcus Autism Center Investigational Device and expert clinical assessment.
  Interventions: Device: Marcus Autism Center Investigational Device

INTERVENTIONS:
Device: Marcus Autism Center Investigational Device — This trial will ascertain whether the binary results of autism or not-autism as determined by the Marcus Autism Center Investigational Device match expert clinical diagnostic opinion. The investigational device is designed to measure visual attention to social information in the environment relative to normative, age-specific benchmarks; these measurements assess presence (primary efficacy outcome) and severity (secondary outcomes) of autism spectrum disorder in 16- to 30-month-old children.

SUMMARY:
This is an outpatient, multicenter, prospective, pivotal, double-blind, within-subject comparison trial of the Marcus Autism Center Investigational Device (MAC-ID) diagnostic procedure relative to the gold-standard (reference standard), current best practice expert clinician diagnosis (ECD) of Autism Spectrum Disorder (ASD) in children 16-30 months of age.

Consecutive pediatric patients from the intended population (i.e. children 16-30 months of age) recruited from pediatric referrals and general advertisements will be the subjects of this trial. All subjects will undergo the MAC-ID diagnostic procedure (test). All subjects will also undergo the current best practice clinical diagnostic procedure, using standardized ASD diagnostic instruments and standardized developmental assessments, to produce the ECD of each child's ASD status (reference/gold standard).

The study consists of a screening phase and diagnostic evaluation phase to assess the validity (sensitivity and specificity), safety, and effectiveness of the MAC-ID when used to diagnose ASD.

Subjects will be enrolled in the trial for a period of 1 day. The trial will be completed in approximately 12 months.

The overall study objective is to assess the safety and effectiveness of the MAC-ID to accurately diagnose ASD (primary analysis), as well as to accurately assess severity of ASD (secondary analysis) in very young pediatric subjects.

The primary endpoints of this study are the diagnostic result from the MAC-ID and the diagnostic results from the ECD evaluation, both of which are either positive or negative for ASD. Each subject will undergo the Social Developmental Testing Device procedure and an examination by a clinical expert in the field of ASD diagnosis; all study center site personnel (including the expert clinicians responsible for the ECD evaluation) will be blinded to MAC-ID results.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to participate in this study:

1. Boys and girls between 16 and 30 months of age
2. Generally healthy with no acute illnesses by physical examination
3. Normal or corrected-to-normal vision, in terms of visual acuity and oculomotor function, sufficient to watch short videos. Adequate hearing to hear material presented in videos
4. Subject and parent can communicate meaningfully in English with the principal investigator and the clinical study site staff
5. Subject's parent or guardian is able to read and understand the informed consent form
6. Parent voluntarily provides written informed consent

Exclusion Criteria:

Any subject who meets any of the exclusion criteria will be excluded from participation in this study:

1. Known genetic disorders (e.g., Fragile X, Williams Syndrome, Tuberous Sclerosis, Muscular Dystrophy, Neurofibromatosis, Down Syndrome)
2. Severe hearing or visual impairment as determined on physical examination (e.g., congenital nystagmus, congenital cataracts, previous diagnosis of severe hearing deficits by otoacoustic emissions or auditory brainstem response)
3. Acute illnesses likely to prevent successful or valid data collection, i.e., conjunctivitis, fever, uncontrolled allergy symptoms, etc.
4. Uncontrolled epilepsy or seizure disorder
5. History or presence of a clinically significant medical disease, or a mental state that might confound the study or be detrimental to the subject as determined by the investigator
6. Acute exacerbations of chronic illnesses likely to prevent successful or valid data collection
7. Receiving therapies that may affect vision, i.e., currently receiving or have received the following therapies within 2 weeks of screening: topiramate, chlorpromazine, thioridazine, prednisone, prednisolone (including ophthalmic solutions and ointments), diphenhydramine, or hydroxyzine; or have received ophthalmic antibiotics within 3 days of screening: tobramycin, ciprofloxacin, gatifloxacin, levofloxacin, moxifloxacin and ofloxacin solutions and/or bacitracin ointment
8. Receiving therapies that may affect the ability to focus attention on the videos, i.e., if on central nervous system (CNS) stimulants, CNS depressants, or anticonvulsants, dose must be stable (same dose for at least 2 weeks).
9. Known allergies or sensitivity to the plastic, leather, or metal components used in the materials of the Social Developmental Testing Device seat
10. Unable or unwilling to sit in a car seat, e.g., child has tantrums on nearly all occasions when placed in a car seat and tantrums do not subside within 5 minutes

Ages: 16 Months to 30 Months | Sex: All
Age Groups: Child
Study Population: Subjects will be recruited on the basis of concern for ASD, including children who a parent, caregiver, or clinician suspects may have ASD as well as children who are not suspected to have an ASD.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Presence of Autism Spectrum Disorder | 1 day
  In a sample of 400, 200 ASD and 200 non-ASD, the investigational device binary determination of ASD versus non-ASD will match the clinician best estimate diagnosis with 70/70 sensitivity and specificity

SECONDARY OUTCOMES:
Social disability index | 1 day
  Using the Autism Diagnostic Observation Schedule, 2nd Edition, does the degree of deviation of visual engagement indicate the severity of autism symptomatology
Verbal Ability Index | 1 day
  Using the verbal domains of the Mullen Scales of Early Learning, does the degree of does the degree of deviation of visual engagement indicate the level of verbal abilities
Nonverbal Ability Index | 1 day
  Using the nonverbal domain of the Mullen Scales of Early Learning, does the degree of does the degree of deviation of visual engagement indicate the level of nonverbal abilities

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Klaiman, PhD, Principal Investigator — Children's Healthcare of Atlanta and Emory University
Locations (6):
- United States (6):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jones W, Klaiman C, Richardson S, Lambha M, Reid M, Hamner T, Beacham C, Lewis P, Paredes J, Edwards L, Marrus N, Constantino JN, Shultz S, Klin A. Development and Replication of Objective Measurements of Social Visual Engagement to Aid in Early Diagnosis and Assessment of Autism. JAMA Netw Open. 2023 Sep 5;6(9):e2330145. doi: 10.1001/jamanetworkopen.2023.30145. PMID 37669054
- [Result] Jones W, Klaiman C, Richardson S, Aoki C, Smith C, Minjarez M, Bernier R, Pedapati E, Bishop S, Ence W, Wainer A, Moriuchi J, Tay SW, Klin A. Eye-Tracking-Based Measurement of Social Visual Engagement Compared With Expert Clinical Diagnosis of Autism. JAMA. 2023 Sep 5;330(9):854-865. doi: 10.1001/jama.2023.13295. PMID 37668621
- See also: EarliPoint Evaluation for Autism Spectrum Disorder — https://www.earlitecdx.com/solutions/